CLINICAL TRIAL: NCT06394960
Title: Factors Predicting Blood Pressure Change Associated With Interscalene Block, Prospective and Observational Study
Brief Title: Factors Predicting Blood Pressure Change With Interscalene Block
Status: Completed | Type: Observational
Sponsor: Konya City Hospital (Other)
Responsible Party: Principal Investigator, Mahmut Sami TUTAR, Associate Professor, Department of Anesthesiology and Reanimation, Konya City Hospital
Other Study IDs: 13.11.2023-22850
Record Dates: First submitted 2024-04-29; First posted 2024-05-01 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Systolic Blood Pressure (20% or Greater Increase)
Keywords: Interscalene Block; Blood Pressure Change; Anterior Scalene Muscle Thickness; Hypertensive Patient

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The primary aim of this study is to identify potential anthropometric features that predict the relationship between the Interscalene Block procedure and changes in blood pressure

DETAILED DESCRIPTION:
This prospective, randomized study will be carried out after obtaining the necessary ethical approval and informed consent from the patients. 110 adult volunteer patients who will undergo ISB for shoulder surgery anesthesia will be included in this study. Evaluation of the patients before ISB and anthropometric measurements before and after Interscalene Block will be performed by an anesthesiologist who is not involved in the study.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-III, elective shoulder surgery will be performed

Exclusion Criteria:

* Presence of advanced renal or hepatic insufficiency, serious respiratory or cardiovascular disease
* History of chronic opioid or benzodiazepine use
* Presence of allergy to the local anesthetic drugs used
* ISB contraindication (such as neurological disorder in the extremity to be operated on, diaphragmatic paralysis in the opposite region of the side where the intervention is planned, infection in the intervention area).
* Presence of high level anxiety
* Patients with a Hospital Anxiety and Depression Scale (HADS) cut-off score of 10 for the anxiety subscale and 7 or higher for the depression subscale

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The participating study center will be Konya City Hospital and the research population will consist of volunteer patients who will undergo elective shoulder surgery under interscalene block.
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2024-05-02 (Actual); Primary Completion 2024-07-10 (Actual); Study Completion 2024-07-20 (Actual)

PRIMARY OUTCOMES:
Our primary aim in this study is to determine possible anthropometric features that will predict the relationship between interscalene block procedure and blood pressure change. | 60 minute
  Various anthropometric measurements (such as "neck diameter", "neck length" and "anterior scalene muscle thickness") may be effective in the spread of the local anesthetic agent during ISB, and these measurements may play a role as a factor in the blood pressure change associated with ISB.

SECONDARY OUTCOMES:
The secondary aim of this study is to reveal the relationship between interscalene block and heart rate. | 60 minute
  Various anthropometric measurements (such as "neck diameter", "neck length" and "anterior scalene muscle thickness") may be effective in the spread of the local anesthetic agent during ISB, and these measurements may play a role as a factor in the heart rate change associated with ISB.

CONTACTS AND LOCATIONS:
Locations (1):
- Konya City Hospital, Konya, Karatay, Turkey (Türkiye)

REFERENCES:
- [Derived] Tutar MS, Polat A, Korkmaz R, Aksoy I, Dogar F, Yildirim A, Satici MH, Yildiz M, Kozanhan B. Prediction of hypertensive responses associated with interscalene block, a prospective cohort study. BMC Anesthesiol. 2025 Feb 19;25(1):82. doi: 10.1186/s12871-025-02947-w. PMID 39972410